CLINICAL TRIAL: NCT04424225
Title: Visual Surround Suppression and Perceptual Expectation Under Psilocybin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Could not secure additional funding to continue the study. Pilot phase of study completed.
Sponsor: University of Minnesota (Other)
Collaborators: Heffter Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PSYCH-2019-28235
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Results first posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Perception Disturbance; Visual Suppression; Psychedelic Experiences
MeSH Terms: interventions — Psilocybin; Niacin; Niacinamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin First (Experimental): Participants in this arm will receive psilocybin first, then niacin
  Interventions: Drug: Psilocybin; Drug: Niacin
- Niacin First (Experimental): Participants in this arm will receive niacin first, then psilocybin
  Interventions: Drug: Psilocybin; Drug: Niacin

INTERVENTIONS:
Drug: Psilocybin — 25 mg capsules (white opaque, Capsugel Vcaps Plus HPMC size 2)
Drug: Niacin — 100 mg capsules (white opaque, Capsugel Vcaps Plus HPMC size 2)
  Other Names: Vitamin B3

SUMMARY:
The prospective pilot study will address the critical need for more precise characterizations of the acute visual effects of the drug psilocybin by measuring the impact of acute psilocybin intoxication on a perceptual task known as visual surround suppression, compared to an active placebo control.

DETAILED DESCRIPTION:
The proposed pilot study will address the critical need for more precise characterizations of the acute visual effects of the drug psilocybin by measuring the impact of acute psilocybin intoxication on a perceptual task known as visual surround suppression, compared to an active placebo control. The data collected in the proposed experiment will make important contributions to knowledge of how psilocybin impacts contextual processing in the brain. Moreover, this will in turn inform the neurobiology of visual surround suppression in general, providing the first investigation of links between surround suppression and serotonergic pathways in humans. Furthermore, the impact of psilocybin on surround suppression will complement recent discoveries of differences in surround suppression present in certain clinical populations. Taken together, these points suggest that this relatively simple and straightforward study could have significant payoff in its contribution to knowledge, not only of the effects of psilocybin but also of key brain processes underpinning human vision and context processing more broadly.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Have at least a high-school level of education or equivalent (e.g. GED), and be able to read and write in English
* General health status: Participants should be in good physical (BMI between 20.0 and 28.0 kg/m2) and psychiatric health.
* Experience taking psilocybin (at the PI's discretion).
* Participants must also have a person that can reliably transport them to and from the CRU for dosing session days.
* Geographic location: Minnesota counties that are approximately within 1 hour driving distance to Twin Cities, including not limited to Hennepin, Ramsey, Washington, Anoka, Wright, Carver, Scott, Dakota, Sherburn
* Participants must be willing to wear a face mask at all times during in-person study visits, except for dosing sessions, to ensure COVID-19 protection.
* Participants must be willing to get a COVID-19 test and share results with the study team prior to all in-person visits.
* Participants must be up-to-date on COVID-19 vaccines, per CDC guidelines, and share a copy of their proof of vaccination status with the study team prior to the consenting visit.
* Agrees to refrain from using recreational drugs while enrolled in the study, including, but not limited to, hallucinogens, ketamine, and marijuana.

Exclusion Criteria:

* Current or past history of meeting DSM-5 criteria for schizophrenia spectrum or other psychotic disorders (except due to another medical condition), or Bipolar I or II Disorder, personality disorder, major depressive disorder, posttraumatic stress disorder, panic disorder, obsessive compulsive disorder, dysthymic disorder.
* Current or past history within the last 5 years of meeting DSM-5 criteria for a moderate or severe alcohol or drug use disorder (excluding caffeine, nicotine, and hallucinogens)
* Those with a first or second-degree relative with a current or past history of meeting DSM-5 criteria for schizophrenia or other psychotic disorders or bipolar I or II disorder, because they might have an underlying genetic susceptibility for psychosis.
* Presence of symptoms of the following DSM-5 disorders within the past 6 months (as assessed by the MINI-7):

  * Major depressive Episode
  * Suicidality
  * Manic and Hypomanic Episodes
  * Panic disorder
  * Agoraphobia
  * Social Anxiety Disorder
  * Obsessive-Compulsive Disorder
  * Posttraumatic Stress Disorder
  * Alcohol Use Disorder
  * Substance Use Disorder (Non-Alcoholic)
  * Psychotic Disorders and Mood Disorders with Psychotic Features
  * Anorexia Nervosa
  * Bulimia Nervosa
  * Binge Eating Disorder
  * Generalized Anxiety Disorder
  * Antisocial Personality Disorder
  * Mood Disorders:
  * Major Depressive Disorder (MDD)
  * MDD with Psychotic Features
  * Bipolar I
  * Bipolar II
  * Other Specified Bipolar and Related Disorder
* Presence of abuse or dependence of drugs measured by the MINI-7 in the past 12 months:

  * Lithium, Sodium Valproate (Depakote), Lamotrigine (Lamictal) - Manic/Bipolar disorders
  * Stimulants: amphetamines, "speed", crystal meth, "crank", Dexedrine, Ritalin, diet pills.
  * Cocaine: snorting, IV, freebase, crack, "speedball".
  * Opiates: heroin, morphine, Dilaudid, opium, Demerol, methadone, Darvon, codeine, Percodan, Vicodin, OxyContin.
  * Dissociative Drugs: PCP (Phencyclidine ,"Angel Dust", "Peace Pill", "Hog"), or ketamine ("Special K").
  * Inhalants: "glue", ethyl chloride, "rush", nitrous oxide ("laughing gas"), amyl or butyl nitrate ("poppers").
  * Cannabis: marijuana, hashish ("hash"), THC, "pot", "grass", "weed", "reefer".
  * Sedatives, Hypnotics or Anxiolytics: Quaalude, Seconal ("reds"), Valium, Xanax, Librium, Ativan, Dalmane, Halcion, barbiturates, Miltown, GHB, Roofinol, "Roofies".
  * Miscellaneous: steroids, nonprescription sleep or diet pills. Cough Medicine?
* History of medication or substance induced psychosis.
* Medically significant condition considered unsuitable for the current study (e.g. diabetes, epilepsy, severe cardiovascular disease, etc)
* History of suicide attempts or mania
* Positive pregnancy test or currently breast-feeding
* Currently taking on a regular (e.g., daily) basis any prescription medications, with the exception of birth control or other hormone therapy
* A strong bias either for or against psychedelic substances, or if their responses about psychedelic use indicate that they abuse them from frequent use (more than once per month, with the exception of microdosing).
* MRI EXCLUSION: we will also exclude anyone with head trauma, claustrophobia incompatible with scanning, cardiac pacemaker, implanted cardiac defibrillator, aneurysm brain clip, inner ear implant, prior history as a metal worker and/or certain metallic objects in the body that cannot be approved for MR scanning by the CMRR safety committee, history of clinically significant vertigo, seizure disorder, middle ear disorder, or double vision, or tattoos that were done less than 4 weeks from the first scheduled MRI.
* Significant movement disorders including tardive dyskinesia that could disrupt EEG recordings will also be excluded.
* Uncontrolled hypertension, with an average blood pressure reading across 4 measurements over 2 separate days greater than 140/90mmHg.
* Unwilling to wear a face mask during in-person study visits that require them.
* Unwilling to get tested for COVID-19 and share results with study personnel prior to all in-person visits.
* Are unvaccinated against COVID-19, are not current with their COVID-19 vaccine booster, or are unwilling to share their proof of COVID-19 vaccination with the study team.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Nielson, PhD, Principal Investigator — University of Minnesota; Link Swanson, PhD(c), Study Director — University of Minnesota; Sophie Jungers, BS, Study Director — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
For data releases, requests for sharing will be made to the PI, Jessica Nielson or the student investigator, Link Swanson, and/or co-investigators Michael-Paul Schallmo, Kathryn Cullen, or Ranji Varghese and granted on an individual basis
URL: https://doi.org/10.17605/OSF.IO/267NH

REFERENCES:
- [Result] Swanson LR, Jungers S, Varghese R, Cullen KR, Evans MD, Nielson JL, Schallmo MP. Enhanced visual contrast suppression during peak psilocybin effects: Psychophysical results from a pilot randomized controlled trial. J Vis. 2024 Nov 4;24(12):5. doi: 10.1167/jov.24.12.5. PMID 39499526
- [Derived] Cotten SW, Strathmann FG, Barrett FS, Labay L, Mullally J, Sherwood AM, Wiegand F. Psychedelics for Medicinal Use: How Will This Alter the Collective Laboratory Consciousness? Clin Chem. 2023 Apr 3;69(4):319-326. doi: 10.1093/clinchem/hvad016. No abstract available. PMID 36881769

RESULTS

PARTICIPANT FLOW:
Groups:
- Psilocybin First, Niacin Second: Participants in this arm will receive psilocybin first, then niacin
  Psilocybin: 25 mg capsules (white opaque, Capsugel Vcaps Plus HPMC size 2)
  Niacin: 100 mg capsules (white opaque, Capsugel Vcaps Plus HPMC size 2)
- Niacin First, Psilocybin Second: Participants in this arm will receive niacin first, then psilocybin
  Psilocybin: 25 mg capsules (white opaque, Capsugel Vcaps Plus HPMC size 2)
  Niacin: 100 mg capsules (white opaque, Capsugel Vcaps Plus HPMC size 2)
Period: Overall Study
Arm/Group | Psilocybin First, Niacin Second | Niacin First, Psilocybin Second
Started | 6 | 4
Completed | 4 | 3
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psilocybin First, Niacin Second | Niacin First, Psilocybin Second | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (9.2) | 34.8 (3.2) | 35.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Psychophysical Descrimination Threshold - No Surround Suppression (NS) Dose 1
Description: No surround suppression condition for visual psychophysics tasks, consisting of perceptual judgments (e.g., subject reported which of two visual stimuli presented appeared to have higher contrast). Based on these responses, psychophysical discrimination thresholds are calculated using an adaptive staircase technique and reported in units of percent contrast.
  .
Time Frame: 3 hours after dose 1
Measure: Mean (Standard Deviation); unit: percent contrast
Groups:
- Psilocybin: Received Psilocybin
- Niacin: Received Niacin
Arm/Group | Psilocybin | Niacin
Number analyzed (Participants) | 3 | 3
percent contrast | .4849 (.11731) | .499 (.04398)

2. Primary Outcome: Psychophysical Descrimination Threshold - No Surround Suppression (NS) Dose 2
Description: as for outcome 1
Time Frame: 3 hours after dose 2
Measure: Mean (Standard Deviation); unit: percent contrast
Arm/Group | Psilocybin | Niacin
Number analyzed (Participants) | 3 | 3
percent contrast | .4756 (.11254) | .4772 (.04711)

3. Primary Outcome: Psychophysical Descrimination Threshold - Orthogonal Surround Suppression (OS) Dose 1
Description: Orthogonal surround suppression condition for visual psychophysics tasks, consisting of perceptual judgments (e.g., subject reported which of two visual stimuli presented appeared to have higher contrast). Based on these responses, psychophysical discrimination thresholds are calculated using an adaptive staircase technique and reported in units of percent contrast. Orthogonal surround suppression condition (OS).
Time Frame: 3 hours after dose 1
Measure: Mean (Standard Deviation); unit: percent contrast
Arm/Group | Psilocybin | Niacin
Number analyzed (Participants) | 3 | 3
percent contrast | .3841 (.17284) | .4491 (.06183)

4. Primary Outcome: Psychophysical Descrimination Threshold - Orthogonal Surround Suppression (OS) Dose 2
Description: as for outcome 3
Time Frame: 3 hours after dose 2
Measure: Mean (Standard Deviation); unit: percent contrast
Arm/Group | Psilocybin | Niacin
Number analyzed (Participants) | 3 | 3
percent contrast | .4678 (.12891) | .4261 (.03799)

5. Primary Outcome: Psychophysical Descrimination Threshold - Parallel Surround Suppression (PS) Dose 1
Description: Parallel surround suppresion condition for visual psychophysics tasks consisting of perceptual judgments (e.g., subject reported which of two visual stimuli presented appeared to have higher contrast). Based on these responses, psychophysical discrimination thresholds are calculated using an adaptive staircase technique and reported in units of percent contrast. Parallel surround suppression condition (PS).
  .
Time Frame: 3 hours after dose 1
Measure: Mean (Standard Deviation); unit: percent contrast
Arm/Group | Psilocybin | Niacin
Number analyzed (Participants) | 3 | 3
percent contrast | .3015 (.18275) | .3988 (.10744)

6. Primary Outcome: Psychophysical Descrimination Threshold - Parallel Surround Suppression (PS) Dose 2
Description: as for outcome 5
Time Frame: 3 hours after dose 2
Measure: Mean (Standard Deviation); unit: percent contrast
Arm/Group | Psilocybin | Niacin
Number analyzed (Participants) | 3 | 3
percent contrast | .4195 (.13829) | .3672 (.06696)

ADVERSE EVENTS:
Time Frame: Week 12
Arm/Group | Psilocybin | Niacin
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 6/9 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psilocybin (N=9) | Niacin (N=8)
BackPain (General disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 4 (7) | 1 (1)
sleep disturbance (General disorders) | 2 (2) | 1 (3)
stomach pain (General disorders) | 2 (2) | 2 (2)
Nausea (General disorders) | 3 (4) | 0 (0)
Emotional (General disorders) | 2 (3) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of funding. Data from primary outcome for psychophysics and secondary analysis for visual event related potentials (vERP) are for the first 6 participants, as part of Dr. Link Swansons dissertation. Raw neuroimaging data will be deposited into OpenNeuro for ongoing data analysis and data sharing with the broader research community.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT04424225/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT04424225/ICF_001.pdf